CLINICAL TRIAL: NCT02977247
Title: ARM 2: A Prospective, Multicenter, Multi-arm, Clinical Case Collection Program to Acquire Breast Image Data and Establish an Image Library of Exams for Use in Future Research Studies, Training, and Product Development Efforts.
Brief Title: Delphinus SoftVue Prospective Case Collection - ARM 2
Acronym: SV PCC ARM2
Status: Completed | Type: Observational
Sponsor: Delphinus Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DMT-2015.001 ARM 2; Protocol ID: 20151525 (Other: Western IRB)
Record Dates: First submitted 2016-11-23; First posted 2016-11-30 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Breast Neoplasms
Keywords: SoftVue; Dense Breast Tissue; Breast Screening; Abnormal Breast; Normal Breast; Breast Imaging; Breast Biopsy; Mammography; Tomosynthesis; Automated Breast Ultrasound; Breast Cancer; Breast Carcinoma; Breast Tumors; Mammary Carcinoma; Malignant Breast Tumor; Mammary Neoplasm; Mammary Cancer; ABUS; AWBUS; Breast Tomography; ATUS; ABTUS; Mammogram; 3D Mammogram; 3D ABUS; 3D Breast Ultrasound; DBT; FFDM; Digital Mammography; Breast Ultrasound; Dense Breasts; Breast Density; Dense Parenchyma; Asymptomatic; Delphinus; Delphinus Medical Technologies; Diagnostic Breast Imaging
MeSH Terms: conditions — Breast Neoplasms; Mammary Neoplasms, Animal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women undergoing routine diagnostic breast evaluation: Non-Interventional: Women presenting to enrollment sites for diagnostic examinations of symptoms or imaging findings, as recommended by a physician, and assigned BI-RADS category 4 or 5 (biopsy indicated).
  Interventions: Other: Non-Interventional; Device: Automated Whole Breast Ultrasound

INTERVENTIONS:
Other: Non-Interventional — Only standard care procedures will be performed for clinical intervention and diagnostic purposes.
  Other Names: Standard Medical Care
Device: Automated Whole Breast Ultrasound — Bilateral breast ultrasound images will be captured, but not clinically evaluated for diagnostic purposes by a physician.
  Other Names: SoftVue, AWBUS, ABUS, 3D Breast Ultrasound, 3D ABUS, 3D Ultrasound, 3D US

SUMMARY:
The SoftVue™ is a whole breast ultrasound system with an automated scanning curvilinear ring-array transducer that employs UST. It is currently cleared under FDA 510(k) K123209 and K142517 for use as both a B-mode ultrasonic breast imaging system and color imaging of transmission data (sound speed and attenuation). SoftVue™ is not intended to be used as a replacement for screening mammography.

SoftVue uses non-ionizing ultrasound energy to generate tomographic image volumes of the whole breast. While the patient lays prone on a padded table with one breast comfortably submerged in a bath of warm water, a ring-shaped transducer, 22 cm in diameter, encircles the breast and pulses low-frequency sound waves through the water and into the breast tissue. More than 2000 elements in the curvilinear transducer's 360 degree array emit and receive ultrasound signals to analyze echoes from the breast anatomy in all directions, from the chest wall to the nipple. Not only does SoftVue capture data from the reflection of the sound waves off of tissue boundaries and structures within the breast, but because the transducer surrounds the whole breast, SoftVue also captures signals that are transmitted through the breast. This additional transmission data enhances the visualization of the anatomic structure of the breast tissue and is not currently available in any other commercially marketed breast ultrasound device.

This prospective, multicenter, multi-arm, clinical case collection program is IRB-approved and will be conducted in compliance with Good Clinical Practice, the Declaration of Helsinki and all applicable regulatory requirements. Arm 2 aims to collectively enroll up to 1,000 women at a total of up to 8 clinical sites. The design of Arm 2 in this protocol is strictly limited to case collection and is non-interventional; any investigational and/or statistical plans for future analyses will be prepared and registered separately, if they are applicable to the requirements of FDAAA 801.

Arm 2 is limited to the cohort of diagnostic female patients of any breast density composition category, who have been recommended for a breast biopsy (BI-RADS 4 or 5) after diagnostic imaging, or who have confirmed imaging findings. Matched sets of diagnostic imaging and SV exams, from the same patient, demographic information, and clinical outcome data, will be collected during diagnostic workup. Ultrasound characteristics for all types of lesions, whether they are benign or malignant, will be collected as well as objective and subjective breast density composition data. Ultrasound image data may be acquired with modified SoftVue devices, which have passed safety and quality evaluations per Delphinus' quality management system (QMS) and satisfy design change control standards, at select clinical sites in accordance with 21 CFR 812.2 (b), as a routine part of feasibility, validation, and verification testing for engineering and product development purposes.

The exams and clinical data accumulated in this prospective case collection (PCC) protocol will populate a database from which future investigations may be designed for peer reviewed publication, development of user training curricula, building teaching case, and creating new marketing materials for SoftVue.

DETAILED DESCRIPTION:
MEDICAL DEVICES:

* SoftVue™ (SV) automated whole breast ultrasound system, 510(k) Cleared for B-Mode ultrasound breast imaging, manufactured by Delphinus Medical Technologies.
* SoftVue™ with device modifications (software, hardware, user-interface), safety-tested for human use to complete feasibility, verification, and validation testing as a routine part of product development and performed in accordance with FDA 21 CFR 812.2 (b), manufactured by Delphinus Medical Technologies.
* Full-field digital mammography (FFDM), FDA Approved for breast screening and diagnosis, various manufacturers. (If clinically indicated)
* Digital breast tomosynthesis (DBT), FDA Approved for breast screening and diagnosis, various manufacturers.
* Handheld Ultrasound (HHUS), FDA-Cleared for diagnostic breast imaging, various manufacturers. (If clinically indicated)
* Other diagnostic tests and medical device examinations of the breast, including, but not limited to MRI, BSGI, PET, biopsy, and elastography, on the order of a licensed physician, when clinically indicated.

OBJECTIVES:

* Primary: To establish a library of cases for use in future SoftVue™ research studies, user training, and marketing.
* Secondary: Determine the frequency and severity of adverse events (AEs) to further evaluate the safety of SoftVue.

ENDPOINTS:

From multiple clinical sites whichever comes first:

• Up to 1,000 total enrolled subjects

SITES:

At least six (≥ 6) qualified clinical sites in the United States

* MQSA Certified
* Digital Breast Tomosynthesis Screening Program Implemented
* Academic, Community Hospital, or Private Practice Setting

PROJECT DESIGN AND PROCEDURES:

* Potential participants will be recruited from the group of women presenting for diagnostic evaluation or biopsy at multiple clinical sites.
* All participants will complete the same standard care diagnostic evaluations that were recommended by a physician
* Eligible patients will receive a SV scan at the time of their scheduled diagnostic appointments, preferably prior to biopsy
* Investigators at the sites will compare SV images to the accompanying diagnostic images and pathology results
* No clinical SV interpretation will be performed and no clinical interventions will be made or changed based on SV images
* All evaluation results, diagnosis and treatment outcomes will be recorded
* Cancer status for all participants will be surveyed from program entry until and including the completion of physician recommended diagnostic workup
* A case will be determined cancer negative if the participant has non-malignant breast biopsy findings or confirmed non-suspicious diagnostic breast imaging findings
* A case will be determined cancer positive if a pathological evaluation confirms a breast cancer diagnosis (malignancy)

STATISTICAL ANALYSIS:

* Demographic characteristics (age, race, and ethnicity) and other baseline characteristics (e.g., project arm, project site, breast density, lesion-specific characteristics) will be tabulated for all participants.
* A flow diagram or table will illustrate patient disposition ("accountability of patient cohort") including reasons for ineligibility and/or unevaluability.
* Safety will be summarized for all enrolled women. With the exception of anticipated events, adverse events (AEs) and serious adverse events (SAEs), occurring from the time of enrollment (SoftVue) and for 24 hours following the conclusion of the SoftVue exam, will be recorded.
* A separate statistical plan will be developed for any future analysis that includes justification of sample size and, if applicable to the requirements of FDAAA 801, will be registered separately in order to share the results.

ELIGIBILITY:
Inclusion Criteria

* Female
* Any race or ethnicity
* Age 18 or older
* Findings of concern on clinical breast exam or imaging
* Scheduled for diagnostic imaging, needle biopsy, excisional biopsy, or post-needle-biopsy visit
* Diagnostic imaging assessment category BI-RADS 4 or 5 and willing to undergo biopsy(ies) or, per the Principal Investigator, subject's case would be beneficial for use in the lesion atlas or teaching library
* Agrees to be contacted by site staff if a recommended biopsy is not completed within the appropriate time frame

Exclusion Criteria

* Unwilling/unable to comply with the protocol and follow-up recommendations
* Lumpectomy or excisional biopsy of the primary region of interest performed prior to SoftVue imaging, such that there are not sufficient findings to make the case useful for the lesion atlas or teaching library
* Weight exceeds 350lbs
* Currently pregnant or lactating by patient self-report
* Weeping rash, open wounds, or unhealed sores on the breast
* Bilateral mastectomy
* Unable to lay prone on the scan table for up to 15 minutes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Arm 2 is limited to the cohort of diagnostic women of any breast density composition category, who have been recommended for a breast biopsy (BI-RADS 4 or 5) after diagnostic imaging. Matched sets of diagnostic imaging with DBT* and SV exams from the same patient, demographic information, and clinical outcome data, will be collected during diagnostic workup. Ultrasound characteristics for all types of lesions, whether they are benign or malignant, will be collected as well as objective and subjective breast density composition data. Ultrasound image data may be acquired with modified SoftVue devices, which have passed safety and quality evaluations per Delphinus' quality management system (QMS) and satisfy design change control standards, at select clinical sites in accordance with 21 CFR 812.2 (b), as a routine part of feasibility, validation, and verification testing for engineering and product development purposes.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
No Breast Cancer | Current Diagnostic Evaluation Episode, 0 to 60 Days
  Non-Cancer cases, confirmed by normal or negative breast imaging findings or concordant breast biopsy with benign pathology.
Breast Cancer | Current Diagnostic Evaluation Episode, 0 to 60 Days
  Cancer cases, confirmed by breast biopsy with malignant pathology

CONTACTS AND LOCATIONS:
Overall Officials: Mary W Yamashita, MD, Principal Investigator — Keck School of Medicine, University of Southern California
Locations (10):
- United States (10):
  - USC Keck School of Medicine, Los Angeles, California
  - Mount Sinai Medical Center, Miami Beach, Florida
  - SouthCoast Imaging, Savannah, Georgia
  - Beaumont Dearborn Breast Care Center, Dearborn, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mercy Imaging Services, Washington, Missouri
  - Elizabeth Wende Breast Care, Rochester, New York
  - UNC Breast Imaging Center, Chapel Hill, North Carolina
  - Weinstein Imaging Associates, Pittsburgh, Pennsylvania
  - Ascension St. Elizabeth, Radiology Associates of the Fox Valley, Appleton, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tabar L, Duffy SW, Vitak B, Chen HH, Prevost TC. The natural history of breast carcinoma: what have we learned from screening? Cancer. 1999 Aug 1;86(3):449-62. PMID 10430253
- [Background] Duffy SW, Tabar L, Chen HH, Holmqvist M, Yen MF, Abdsalah S, Epstein B, Frodis E, Ljungberg E, Hedborg-Melander C, Sundbom A, Tholin M, Wiege M, Akerlund A, Wu HM, Tung TS, Chiu YH, Chiu CP, Huang CC, Smith RA, Rosen M, Stenbeck M, Holmberg L. The impact of organized mammography service screening on breast carcinoma mortality in seven Swedish counties. Cancer. 2002 Aug 1;95(3):458-69. doi: 10.1002/cncr.10765. PMID 12209737
- [Background] Duffy SW, Smith RA, Gabe R, Tabar L, Yen AM, Chen TH. Screening for breast cancer. Surg Oncol Clin N Am. 2005 Oct;14(4):671-97. doi: 10.1016/j.soc.2005.06.001. PMID 16226686
- [Background] Paci E, Duffy SW, Giorgi D, Zappa M, Crocetti E, Vezzosi V, Bianchi S, del Turco MR. Quantification of the effect of mammographic screening on fatal breast cancers: The Florence Programme 1990-96. Br J Cancer. 2002 Jul 1;87(1):65-9. doi: 10.1038/sj.bjc.6600301. PMID 12085258
- [Background] Tabar L, Duffy SW, Yen MF, Warwick J, Vitak B, Chen HH, Smith RA. All-cause mortality among breast cancer patients in a screening trial: support for breast cancer mortality as an end point. J Med Screen. 2002;9(4):159-62. doi: 10.1136/jms.9.4.159. PMID 12518005
- [Background] Swedish Organised Service Screening Evaluation Group. Effect of mammographic service screening on stage at presentation of breast cancers in Sweden. Cancer. 2007 Jun 1;109(11):2205-12. doi: 10.1002/cncr.22671. PMID 17471486
- [Background] Swedish Organised Service Screening Evaluation Group. Reduction in breast cancer mortality from organized service screening with mammography: 1. Further confirmation with extended data. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):45-51. doi: 10.1158/1055-9965.EPI-05-0349. PMID 16434585
- [Background] Swedish Organised Service Screening Evaluation Group. Reduction in breast cancer mortality from the organised service screening with mammography: 2. Validation with alternative analytic methods. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):52-6. doi: 10.1158/1055-9965.EPI-05-0953. PMID 16434586
- [Background] Hakama M, Pukkala E, Heikkila M, Kallio M. Effectiveness of the public health policy for breast cancer screening in Finland: population based cohort study. BMJ. 1997 Mar 22;314(7084):864-7. doi: 10.1136/bmj.314.7084.864. PMID 9093096
- [Background] Tabar L, Vitak B, Chen TH, Yen AM, Cohen A, Tot T, Chiu SY, Chen SL, Fann JC, Rosell J, Fohlin H, Smith RA, Duffy SW. Swedish two-county trial: impact of mammographic screening on breast cancer mortality during 3 decades. Radiology. 2011 Sep;260(3):658-63. doi: 10.1148/radiol.11110469. Epub 2011 Jun 28. PMID 21712474
- [Background] Michaelson JS, Silverstein M, Wyatt J, Weber G, Moore R, Halpern E, Kopans DB, Hughes K. Predicting the survival of patients with breast carcinoma using tumor size. Cancer. 2002 Aug 15;95(4):713-23. doi: 10.1002/cncr.10742. PMID 12209713
- [Background] Smith RA, Duffy SW, Gabe R, Tabar L, Yen AM, Chen TH. The randomized trials of breast cancer screening: what have we learned? Radiol Clin North Am. 2004 Sep;42(5):793-806, v. doi: 10.1016/j.rcl.2004.06.014. PMID 15337416
- [Background] Kolb TM, Lichy J, Newhouse JH. Comparison of the performance of screening mammography, physical examination, and breast US and evaluation of factors that influence them: an analysis of 27,825 patient evaluations. Radiology. 2002 Oct;225(1):165-75. doi: 10.1148/radiol.2251011667. PMID 12355001
- [Background] Kerlikowske K, Grady D, Barclay J, Sickles EA, Ernster V. Effect of age, breast density, and family history on the sensitivity of first screening mammography. JAMA. 1996 Jul 3;276(1):33-8. PMID 8667536
- [Background] Pisano ED, Gatsonis C, Hendrick E, Yaffe M, Baum JK, Acharyya S, Conant EF, Fajardo LL, Bassett L, D'Orsi C, Jong R, Rebner M; Digital Mammographic Imaging Screening Trial (DMIST) Investigators Group. Diagnostic performance of digital versus film mammography for breast-cancer screening. N Engl J Med. 2005 Oct 27;353(17):1773-83. doi: 10.1056/NEJMoa052911. Epub 2005 Sep 16. PMID 16169887
- [Background] Cole EB, Pisano ED, Kistner EO, Muller KE, Brown ME, Feig SA, Jong RA, Maidment AD, Staiger MJ, Kuzmiak CM, Freimanis RI, Lesko N, Rosen EL, Walsh R, Williford M, Braeuning MP. Diagnostic accuracy of digital mammography in patients with dense breasts who underwent problem-solving mammography: effects of image processing and lesion type. Radiology. 2003 Jan;226(1):153-60. doi: 10.1148/radiol.2261012024. PMID 12511684
- [Background] Haas BM, Kalra V, Geisel J, Raghu M, Durand M, Philpotts LE. Comparison of tomosynthesis plus digital mammography and digital mammography alone for breast cancer screening. Radiology. 2013 Dec;269(3):694-700. doi: 10.1148/radiol.13130307. Epub 2013 Oct 28. PMID 23901124
- [Background] Svahn TM, Chakraborty DP, Ikeda D, Zackrisson S, Do Y, Mattsson S, Andersson I. Breast tomosynthesis and digital mammography: a comparison of diagnostic accuracy. Br J Radiol. 2012 Nov;85(1019):e1074-82. doi: 10.1259/bjr/53282892. Epub 2012 Jun 6. PMID 22674710
- [Background] Rafferty EA, Park JM, Philpotts LE, Poplack SP, Sumkin JH, Halpern EF, Niklason LT. Assessing radiologist performance using combined digital mammography and breast tomosynthesis compared with digital mammography alone: results of a multicenter, multireader trial. Radiology. 2013 Jan;266(1):104-13. doi: 10.1148/radiol.12120674. Epub 2012 Nov 20. PMID 23169790
- [Background] Wolfe JN. Breast patterns as an index of risk for developing breast cancer. AJR Am J Roentgenol. 1976 Jun;126(6):1130-7. doi: 10.2214/ajr.126.6.1130. PMID 179369
- [Background] Ursin G, Hovanessian-Larsen L, Parisky YR, Pike MC, Wu AH. Greatly increased occurrence of breast cancers in areas of mammographically dense tissue. Breast Cancer Res. 2005;7(5):R605-8. doi: 10.1186/bcr1260. Epub 2005 Jun 8. PMID 16168104
- [Background] Titus-Ernstoff L, Tosteson AN, Kasales C, Weiss J, Goodrich M, Hatch EE, Carney PA. Breast cancer risk factors in relation to breast density (United States). Cancer Causes Control. 2006 Dec;17(10):1281-90. doi: 10.1007/s10552-006-0071-1. PMID 17111260
- [Background] Boyd NF, Guo H, Martin LJ, Sun L, Stone J, Fishell E, Jong RA, Hislop G, Chiarelli A, Minkin S, Yaffe MJ. Mammographic density and the risk and detection of breast cancer. N Engl J Med. 2007 Jan 18;356(3):227-36. doi: 10.1056/NEJMoa062790. PMID 17229950
- [Background] Boyd NF, Martin LJ, Yaffe MJ, Minkin S. Mammographic density: a hormonally responsive risk factor for breast cancer. J Br Menopause Soc. 2006 Dec;12(4):186-93. doi: 10.1258/136218006779160436. PMID 17178021
- [Background] Torres-Mejia G, De Stavola B, Allen DS, Perez-Gavilan JJ, Ferreira JM, Fentiman IS, Dos Santos Silva I. Mammographic features and subsequent risk of breast cancer: a comparison of qualitative and quantitative evaluations in the Guernsey prospective studies. Cancer Epidemiol Biomarkers Prev. 2005 May;14(5):1052-9. doi: 10.1158/1055-9965.EPI-04-0717. PMID 15894652
- [Background] Stone J, Dite GS, Gunasekara A, English DR, McCredie MR, Giles GG, Cawson JN, Hegele RA, Chiarelli AM, Yaffe MJ, Boyd NF, Hopper JL. The heritability of mammographically dense and nondense breast tissue. Cancer Epidemiol Biomarkers Prev. 2006 Apr;15(4):612-7. doi: 10.1158/1055-9965.EPI-05-0127. PMID 16614099
- [Background] Kolb TM, Lichy J, Newhouse JH. Occult cancer in women with dense breasts: detection with screening US--diagnostic yield and tumor characteristics. Radiology. 1998 Apr;207(1):191-9. doi: 10.1148/radiology.207.1.9530316.
- [Background] Checka CM, Chun JE, Schnabel FR, Lee J, Toth H. The relationship of mammographic density and age: implications for breast cancer screening. AJR Am J Roentgenol. 2012 Mar;198(3):W292-5. doi: 10.2214/AJR.10.6049. PMID 22358028
- [Background] Sprague BL, Gangnon RE, Burt V, Trentham-Dietz A, Hampton JM, Wellman RD, Kerlikowske K, Miglioretti DL. Prevalence of mammographically dense breasts in the United States. J Natl Cancer Inst. 2014 Sep 12;106(10):dju255. doi: 10.1093/jnci/dju255. Print 2014 Oct. PMID 25217577
- [Background] Rieber A, Brambs HJ, Gabelmann A, Heilmann V, Kreienberg R, Kuhn T. Breast MRI for monitoring response of primary breast cancer to neo-adjuvant chemotherapy. Eur Radiol. 2002 Jul;12(7):1711-9. doi: 10.1007/s00330-001-1233-x. Epub 2002 Feb 14. PMID 12111062
- [Background] King V, Brooks JD, Bernstein JL, Reiner AS, Pike MC, Morris EA. Background parenchymal enhancement at breast MR imaging and breast cancer risk. Radiology. 2011 Jul;260(1):50-60. doi: 10.1148/radiol.11102156. Epub 2011 Apr 14. PMID 21493794
- [Background] Saslow D, Boetes C, Burke W, Harms S, Leach MO, Lehman CD, Morris E, Pisano E, Schnall M, Sener S, Smith RA, Warner E, Yaffe M, Andrews KS, Russell CA; American Cancer Society Breast Cancer Advisory Group. American Cancer Society guidelines for breast screening with MRI as an adjunct to mammography. CA Cancer J Clin. 2007 Mar-Apr;57(2):75-89. doi: 10.3322/canjclin.57.2.75. PMID 17392385
- [Background] Kuhl CK, Schrading S, Strobel K, Schild HH, Hilgers RD, Bieling HB. Abbreviated breast magnetic resonance imaging (MRI): first postcontrast subtracted images and maximum-intensity projection-a novel approach to breast cancer screening with MRI. J Clin Oncol. 2014 Aug 1;32(22):2304-10. doi: 10.1200/JCO.2013.52.5386. Epub 2014 Jun 23. PMID 24958821
- [Background] Corsetti V, Ferrari A, Ghirardi M, Bergonzini R, Bellarosa S, Angelini O, Bani C, Ciatto S. Role of ultrasonography in detecting mammographically occult breast carcinoma in women with dense breasts. Radiol Med. 2006 Apr;111(3):440-8. doi: 10.1007/s11547-006-0040-5. Epub 2006 Apr 11. English, Italian. PMID 16683089
- [Background] Crystal P, Strano SD, Shcharynski S, Koretz MJ. Using sonography to screen women with mammographically dense breasts. AJR Am J Roentgenol. 2003 Jul;181(1):177-82. doi: 10.2214/ajr.181.1.1810177. PMID 12818853
- [Background] Berg WA, Zhang Z, Lehrer D, Jong RA, Pisano ED, Barr RG, Bohm-Velez M, Mahoney MC, Evans WP 3rd, Larsen LH, Morton MJ, Mendelson EB, Farria DM, Cormack JB, Marques HS, Adams A, Yeh NM, Gabrielli G; ACRIN 6666 Investigators. Detection of breast cancer with addition of annual screening ultrasound or a single screening MRI to mammography in women with elevated breast cancer risk. JAMA. 2012 Apr 4;307(13):1394-404. doi: 10.1001/jama.2012.388. PMID 22474203
- [Background] Hooley RJ, Greenberg KL, Stackhouse RM, Geisel JL, Butler RS, Philpotts LE. Screening US in patients with mammographically dense breasts: initial experience with Connecticut Public Act 09-41. Radiology. 2012 Oct;265(1):59-69. doi: 10.1148/radiol.12120621. Epub 2012 Jun 21. PMID 22723501
- [Background] Kelly KM, Dean J, Comulada WS, Lee SJ. Breast cancer detection using automated whole breast ultrasound and mammography in radiographically dense breasts. Eur Radiol. 2010 Mar;20(3):734-42. doi: 10.1007/s00330-009-1588-y. Epub 2009 Sep 2. PMID 19727744
- [Background] Corsetti V, Houssami N, Ferrari A, Ghirardi M, Bellarosa S, Angelini O, Bani C, Sardo P, Remida G, Galligioni E, Ciatto S. Breast screening with ultrasound in women with mammography-negative dense breasts: evidence on incremental cancer detection and false positives, and associated cost. Eur J Cancer. 2008 Mar;44(4):539-44. doi: 10.1016/j.ejca.2008.01.009. Epub 2008 Feb 11. PMID 18267357
- [Background] Leconte I, Feger C, Galant C, Berliere M, Berg BV, D'Hoore W, Maldague B. Mammography and subsequent whole-breast sonography of nonpalpable breast cancers: the importance of radiologic breast density. AJR Am J Roentgenol. 2003 Jun;180(6):1675-9. doi: 10.2214/ajr.180.6.1801675. PMID 12760942
- [Background] Kaplan SS. Clinical utility of bilateral whole-breast US in the evaluation of women with dense breast tissue. Radiology. 2001 Dec;221(3):641-9. doi: 10.1148/radiol.2213010364. PMID 11719658
- [Background] Buchberger W, Niehoff A, Obrist P, DeKoekkoek-Doll P, Dunser M. Clinically and mammographically occult breast lesions: detection and classification with high-resolution sonography. Semin Ultrasound CT MR. 2000 Aug;21(4):325-36. doi: 10.1016/s0887-2171(00)90027-1. PMID 11014255
- [Background] Gordon PB, Goldenberg SL. Malignant breast masses detected only by ultrasound. A retrospective review. Cancer. 1995 Aug 15;76(4):626-30. doi: 10.1002/1097-0142(19950815)76:43.0.co;2-z. PMID 8625156
- [Background] Berg WA, Blume JD, Cormack JB, Mendelson EB, Lehrer D, Bohm-Velez M, Pisano ED, Jong RA, Evans WP, Morton MJ, Mahoney MC, Larsen LH, Barr RG, Farria DM, Marques HS, Boparai K; ACRIN 6666 Investigators. Combined screening with ultrasound and mammography vs mammography alone in women at elevated risk of breast cancer. JAMA. 2008 May 14;299(18):2151-63. doi: 10.1001/jama.299.18.2151. PMID 18477782
- [Background] Berg WA, Blume JD, Cormack JB, Mendelson EB. Operator dependence of physician-performed whole-breast US: lesion detection and characterization. Radiology. 2006 Nov;241(2):355-65. doi: 10.1148/radiol.2412051710. PMID 17057064
- [Background] Brem RF, Tabar L, Duffy SW, Inciardi MF, Guingrich JA, Hashimoto BE, Lander MR, Lapidus RL, Peterson MK, Rapelyea JA, Roux S, Schilling KJ, Shah BA, Torrente J, Wynn RT, Miller DP. Assessing improvement in detection of breast cancer with three-dimensional automated breast US in women with dense breast tissue: the SomoInsight Study. Radiology. 2015 Mar;274(3):663-73. doi: 10.1148/radiol.14132832. Epub 2014 Oct 17. PMID 25329763
- [Background] Ranger B, Littrup PJ, Duric N, Chandiwala-Mody P, Li C, Schmidt S, Lupinacci J. Breast ultrasound tomography versus MRI for clinical display of anatomy and tumor rendering: preliminary results. AJR Am J Roentgenol. 2012 Jan;198(1):233-9. doi: 10.2214/AJR.11.6910. PMID 22194502
- [Background] Mandelson MT, Oestreicher N, Porter PL, White D, Finder CA, Taplin SH, White E. Breast density as a predictor of mammographic detection: comparison of interval- and screen-detected cancers. J Natl Cancer Inst. 2000 Jul 5;92(13):1081-7. doi: 10.1093/jnci/92.13.1081. PMID 10880551
- [Background] Houssami N, Irwig L, Ciatto S. Radiological surveillance of interval breast cancers in screening programmes. Lancet Oncol. 2006 Mar;7(3):259-65. doi: 10.1016/S1470-2045(06)70617-9. PMID 16510335
- [Background] Roubidoux MA, Bailey JE, Wray LA, Helvie MA. Invasive cancers detected after breast cancer screening yielded a negative result: relationship of mammographic density to tumor prognostic factors. Radiology. 2004 Jan;230(1):42-8. doi: 10.1148/radiol.2301020589. PMID 14695385
- See also: Delphinus Medical Technologies — https://www.delphinusmt.com/